CLINICAL TRIAL: NCT05159297
Title: Normative Reference Values of Sideways Walking, Tandem Walking, Cross-stepping, Heel Walking and Toe Walking Among Children
Brief Title: Normative Reference Values of Equilibrium Coordination Test Among Children
Status: Completed | Type: Observational
Sponsor: Asir John Samuel (Other)
Collaborators: Maharishi Markandeshwar International School, Mullana (Unknown)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Other Study IDs: MMDU/IEC/2153; U1111-1269-9876 (Other: Universal Trial Number (WHO))
Record Dates: First submitted 2021-10-01; First posted 2021-12-16 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Coordination Disorder, Developmental
Keywords: children; coordination; normal range; postural balance; walking
MeSH Terms: conditions — Motor Skills Disorders | interventions — Reference Values

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Reference values — Normative reference values of coordination tests will be obtained

SUMMARY:
A cross-sectional study will be conducted recruiting children of age group 8-15 years. Pilot study has been conducted for the determination of the sample size. The calculated sample size has come out to be, n=378 which can be taken for males and females separately. Stratified random sampling will be done according to age. Child will be asked to perform all tests one by one and the time taken (in seconds) will be noted required to perform the tests. The mean of three readings will be obtained using a mobile-based stop watch.

DETAILED DESCRIPTION:
756 children will be recruited of age group 8-15 years. Five equilibrium coordination tests i.e. Sideways walking, tandem walking, cross-stepping, heel walking and toe walking will be performed by each child and three readings will be recorded. Mean of three readings will be considered as normative reference value of each test respectively.

ELIGIBILITY:
Inclusion Criteria:

* Typically developing school-going children with age group between 8 and 15 years
* Both male and female
* Able to walk independently
* Able to follow verbal commands

Exclusion Criteria:

* Any fracture of lower limb in last 6 months
* Any congenital anomaly affecting lower limb
* Any developmental disorder
* Any open wounds
* Those who are using any kind of assistive devices
* Any condition that affect the health status of the participants during the study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Normal healthy children of age group between 8 and 17 years was recruited
Sampling Method: Probability Sample
Enrollment: 1104 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-09-16 (Actual)

PRIMARY OUTCOMES:
Sideways walking | Immediately after the sideways walking
  This test will be used to find the normative values of sideways walking
Tandem walking | Immediately after the Tandem walking
  This test will be used to find the normative values of tandem walking
Cross stepping | Immediately after the Cross stepping
  This test will be used to find the normative values of cross stepping
Heel Walking | Immediately after the Heel Walking
  This test will be used to find the normative values of heel walking
Toe walking | Immediately after the Toe walking
  This test will be used to find the normative values of toe walking

CONTACTS AND LOCATIONS:
Overall Officials: Nidhi Sharma, PhD Scholar, Principal Investigator — Maharishi Markendeshwar University (Deemed to be University)
Locations (1):
- Maharishi Markandeshwar International School, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aylar MF, Dionisio VC, Jafarnezhadgero A, Parikhani AZ. Body coordination during sit-to-stand in blind and sighted female children. J Biomech. 2020 May 7;104:109708. doi: 10.1016/j.jbiomech.2020.109708. Epub 2020 Feb 28. PMID 32173035
- [Background] Riquelme I, Arnould C, Hatem SM, Bleyenheuft Y. The Two-Arm Coordination Test: Maturation of Bimanual Coordination in Typically Developing Children and Deficits in Children with Unilateral Cerebral Palsy. Dev Neurorehabil. 2019 Jul;22(5):312-320. doi: 10.1080/17518423.2018.1498552. Epub 2018 Jul 19. PMID 30024779
- [Background] McKay MJ, Baldwin JN, Ferreira P, Simic M, Vanicek N, Burns J; 1000 Norms Project Consortium. Normative reference values for strength and flexibility of 1,000 children and adults. Neurology. 2017 Jan 3;88(1):36-43. doi: 10.1212/WNL.0000000000003466. Epub 2016 Nov 23. PMID 27881628
- [Background] Bolk J, Farooqi A, Hafstrom M, Aden U, Serenius F. Developmental Coordination Disorder and Its Association With Developmental Comorbidities at 6.5 Years in Apparently Healthy Children Born Extremely Preterm. JAMA Pediatr. 2018 Aug 1;172(8):765-774. doi: 10.1001/jamapediatrics.2018.1394. PMID 29868837
- [Background] Dunsky A. The Effect of Balance and Coordination Exercises on Quality of Life in Older Adults: A Mini-Review. Front Aging Neurosci. 2019 Nov 15;11:318. doi: 10.3389/fnagi.2019.00318. eCollection 2019. PMID 31803048
- [Background] Lanzino DJ, Rabinstein A, Kinlaw D, Hepburn SB, Ness BM, Olson KJ, Sobie SM, Hollman JH. Coordination tests in persons with acute central nervous system pathology: assessment of interrater reliability and known-group validity. J Neurol Phys Ther. 2012 Sep;36(3):122-30. doi: 10.1097/NPT.0b013e3182641d36. PMID 22850331